CLINICAL TRIAL: NCT04364685
Title: Effect of Walking on Sand With Dietary Intervention in Overweight Type 2 Diabetes Mellitus Patients: A Randomized Controlled Trial.
Brief Title: Effect of Walking on Sand With Dietary Intervention in Overweight Type 2 Diabetes Mellitus Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Majmaah University (Other)
Responsible Party: Principal Investigator, faizan kashoo, PT, Lecturer, Majmaah University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MajmaahUNI
Record Dates: First submitted 2020-04-23; First posted 2020-04-28 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Walking, Difficulty; Diabetes Mellitus, Type 2; Hemoglobin; Hb-SC
MeSH Terms: conditions — Mobility Limitation; Diabetes Mellitus, Type 2; Hemoglobin SC Disease

STUDY DESIGN:
Intervention Model Description: The study consists of two groups, one control group (Normal Walking) and experimental group (sand walking).
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigator responsible for evaluation of patient was blinded to the allocation of the participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal Walking (Active Comparator): The participants performed 30 minutes on levelled surface on the track and field ground. Participants performed moderate intensity walking, self paced.
  Interventions: Other: Walking on Levelled Surface
- Sand Walking (Experimental): The participants performed supervised walking on sand on the 20 meters pathway containing soft sand.The walking on sand for 30 minutes.
  Interventions: Other: Walking on soft-sand

INTERVENTIONS:
Other: Walking on soft-sand — The participants are required to walking on sand for 30 minutes. Walking is self-paced.
  Arms: Sand Walking
Other: Walking on Levelled Surface — The Participants will be require to walk on the firm surface for 30 minutes. The participants would decide the pace of walking.
  Arms: Normal Walking

SUMMARY:
Type 2 Diabetes Meletus(T2DM) is a global health concern. The incidence of T2DM globally is increasing exponentially partly due to unhealthy food habits and sedentary life style.exercise and nutritional intervention is long being reported to improve glycemic control and improve quality of life among individuals with T2DM.

Moderate intensity of walking for 30 minutes is proven to regulate good metabolic control. however, in over weight elderly individuals, joint pain or arthritis walking be a challenging task. therefore, walking on sand which is reported to be easy on joints would be a alternative for those patients.

DETAILED DESCRIPTION:
Uncontrolled T2DM has shown to cause multiple complications and alter the normal physiological process of the body. Prompt dietary management and regular exercises are reported to improve blood glucose homeostasis and eventually improve the quality of life. Physical activity such as regular walking is associated with multiple physical and psychological benefits. Walking and a healthy diet is a cornerstone in the treatment of T2DM. Several studies have shown positive short-term effects of walking in T2DM. Combination of walking and weight training is reported to cause cardiovascular adaptations, muscle hypertrophy, increased capillary density in the muscles of patients with T2DM as well as in healthy people. Furthermore, 30 minutes of brisk walking has shown to improve blood glycemic metabolism and reduces cardiovascular risk factors, such as high blood pressure, lipid disorders, and fat mass buildup. However, the elderly with mild to moderate arthritic changes especially in knee joints make walking a bit more challenging. Sand walking would be the best alternative than firm surface walking with less joint reaction forces. To the best of our knowledge, scientific literature lacks evidence about the effect of sand walking combined with individualized dietary intervention in T2DM. Therefore, the purpose of this study was to compare the effect of sand walking as compared to normal walking on glycemic metabolism, weight, and quality of life in T2DM. The Investigators hypothesize that SW would result in better health benefits than NW in T2DM.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with Type 2 Diabetes for past 1 year.
2. HbA1c between 7-10%.
3. BMI between 25-29.9
4. Age Between 45-75
5. Sedentary

Exclusion Criteria:

1. Diabetic Neuropathy
2. Active Smoker
3. Musculoskeletal conditions
4. Cardiovascular conditions

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2017-01-25 (Actual); Primary Completion 2019-09-26 (Actual); Study Completion 2019-09-28 (Actual)

PRIMARY OUTCOMES:
HbA1c | 16 weeks
  Percentage of hemoglobin A1c

SECONDARY OUTCOMES:
BMI | 16 weeks
  Body mass index
Waist Circumference | 2 years
  the waist circumference was measured by inch tape at the level of Anterior superior iliac spine.
Quality of life-39 | 16 weeks
  The Validated quality of life for diabetes containing 39 items and scoring on a 1-7 Likert scale.

CONTACTS AND LOCATIONS:
Locations (1):
- King Khalid Hospital, Al Majma'ah, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided
The complete data set will be send upon request.